CLINICAL TRIAL: NCT00534222
Title: Unraveling the Relation of Patient's Profile and Therapeutical Effects of Atypicals, Including Quetiapine Effect
Acronym: UPTAQE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-NNL-SER-2005/1; NL 401241 (Registry Identifier: NIS)
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2009-04

CONDITIONS: Mania; Schizophrenia
Keywords: Patients with a manic episode; Patients diagnosed w/schizophrenia, who start a treatment with an atypical antipsychotic & who are at least scored as moderately ill on the CGI at baseline
MeSH Terms: conditions — Mania; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Quetiapine
- Olanzapine
- Risperidone

SUMMARY:
With this observational study we want to examine if the intensity of agitation, the intensity of psychotic symptoms and the presence of sleeping disorder predict the success of the treatment with a atypical antipsychotic after 12 weeks of treatment with patients with a psychotic and/or manic episode. In this study it will be examined what the percentage of patients with a 2-point improvement at the CGI-scale is. Of these group, the responders, retrospective the profile of the responders will be analysed (key-factors and confounders).

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a manic episode or patients diagnosed with schizophrenia (psychotic episode)
* Patients who start a treatment with an atypical antipsychotic : quetiapine, olanzapine or risperidone
* Patients who are prepared to consent to make the coded data available to AstraZeneca
* Patients with a CGI ≥ 4

Exclusion Criteria:

* Patients with a serious underlying disease (including renal or hepatic insufficiency, cancer, cardiovascular diseases and suchlike).
* Contra-indications for quetiapine, olanzapine or risperidone according to the SmPC for these products
* Patients unable to give informed consent according to the attending physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatrist' patients
Sampling Method: Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2005-09; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — AstraZeneca
Locations (6):
- Netherlands (6):
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Alphen Aan de Rigjn
  - Research Site, Amersfoort
  - Research Site, Amstelveen
  - Research Site, Amsterdam